CLINICAL TRIAL: NCT02297035
Title: Linguistic, Anatomic/Metabolic and Biologic Characterisation of the Three Main Variants of Primary Progressive Aphasia : Towards the Rationale for Drug Trials and Specific Language Rehabilitations
Brief Title: Characterisation of Primary Progressives Aphasias
Acronym: CAPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P100137
Record Dates: First submitted 2014-10-10; First posted 2014-11-21 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-02

CONDITIONS: Aphasia Primary Progressive
MeSH Terms: conditions — Pick Disease of the Brain | interventions — Neuroimaging; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PPA patients (Experimental): Experimental (Patients responding to current diagnostic criteria for Primary Progressive Aphasia (PPA) patients) : Behavioural testing, Brain imaging (MRI, PET), Genetic screening (APOE, Progranulin)
  Interventions: Behavioral: Behavioural testing; Other: Brain imaging; Genetic: Genetic screening
- healthy controls (Experimental): Healthy controls : Behavioural testing, Brain imaging (MRI, PET).
  Interventions: Behavioral: Behavioural testing; Other: Brain imaging

INTERVENTIONS:
Behavioral: Behavioural testing
Other: Brain imaging — MRI, PET
Genetic: Genetic screening — APOE, Progranulin
  Arms: PPA patients

SUMMARY:
Primary progressive aphasias (PPA) represent a challenging group of degenerative language diseases that has led to growing interest in the scientific and medical community. However, a full-blown cognitive/linguistic, anatomic and biologic characterization of the three main variants remains incomplete given that the available data derive from relatively small patient samples. Such a three-fold characterisation will be an major milestone with the prospective of providing the rationale for therapeutic interventions comprising specific rehabilitations protocols and pharmacological trials.

The present study addresses theses issues in the three PPA main variants through a cross-sectional and longitudinal investigation exploring 1) cognitive/linguistic features, 2) anatomic/metabolic specifications (MRI-VBM, MRI-fiber tracking, functional connectivity - MRI resting state, PET), and 3) biologic aspects (CSF biomarkers, genetic screening).

DETAILED DESCRIPTION:
Rationale Primary progressive aphasia (PPA) is an umbrella term which identifies a group of neurodegenerative diseases characterized by language deficits. By definition, language disorders are isolated for at least two years; subsequently the disease extends to other cognitive areas leading to a global dementia. Usually PPA affects relatively young patients between 50 and 65 years of age. The outcome is fatal after 10 to 15 years. No treatment is currently available. Three variants of PPA have been described: progressive nonfluent aphasia (PNFA), fluent PPA or semantic dementia (SD), and logopenic progressive aphasia (LPA). These variants are characterized by differences in the nature of the language deficits, the patterns of brain atrophy and the underlying pathology, comprising Alzheimer's pathology in about 30% of patients with PPA . In spite of the growing interest, the cognitive, anatomic and biologic characterization of the 3 PPA variants remains incomplete and the available data derive from studies on small patient samples. However, such a three-fold characterisation is essential in order to provide the rationale for therapeutic interventions comprising both specific rehabilitation of language and pharmacological treatments. In particular, the pharmacological approach crucially depends on a better knowledge of the underlying histopathology (e.g., the existence of Alzheimer pathology), as well as on the understanding of the damaged neural networks that may provide evidence for the implication of specific neurotransmitters. Our aim is to address these issues through exploring a large population of patients with PPA associating psycholinguistic tools, cutting-edge techniques of neuroimaging, CSF biomarker analyses and genetic screening. The study will provide a cross-sectional and longitudinal assessment of PPA patients involving 17 memory centres qualified in the domain of PPA.

Main objective Providing an comprehensive characterisation of the 3 PPA variants through a cross-sectional and longitudinal approach investigating 1) the cognitive features (psycholinguistic), 2) the anatomic/metabolic substrates (structural MRI, DTI-based tractography, functional connectivity - resting state, 18FDG-PET), and 3) the biologic aspects (CSF biomarkers [amyloid-β and tau], genetic screening for mutations in the progranulin gene, apolipoprotein E genotyping).

Secondary objectives

1) Identification of prognostic markers (linguistic, anatomical/metabolic, biologic) for each PPA variant. 2) Identification of predictive markers (linguistic, neuroimaging) for the underlying histopathology (correlation analyses among linguistic, imaging, CSF and genetic markers). 3) Validation of the diagnostic criteria of semantic dementia to distinguish the fluent/semantic variant of PPA and forms with multimodal disorders of semantics (verbal and visual).

Perspectives Providing the rationale for drug trials and for specific language rehabilitations.

Methodology One hundred twenty-five PPA patients and 40 healthy age-matched controls will be included in the study. Patients will be recruited from a national network including the "national center of reference for rare dementias" and 10 associated "Centers of competence" , as well as six additional hospitals, all experienced in the domain of PPA.

Study design: The duration of the study will be three years (18 months inclusion, 18 months exploration). Participants will be assessed at inclusion (M0), at 9 months (M9) and at 18 months (M18). The explorations will be subdivided into 3 work packages, each coordinated by a supervisor. 1) Cognitive work package (M0, M9, M18): A) Neuropsychological and language testing using standardized and internationally validated batteries; B) Neuropsychological battery specially conceived to explore verbal and visual semantics (validation of the new diagnostic criteria of semantic dementia; secondary objective N° 3); C) Language assessment using specifically targeted paradigms based on psycholinguistic models. Imaging work package (M0, M18): A) MRI and MRI-based tractography to detect and quantify cortical atrophy, the involvement of white matter tracts and to study the functional connectivity (resting state fMRI); B) 18FDG-PET to study metabolic defects of the cortex and the basal ganglia. 3) Biologic work package (M0; no controls): Lumbar puncture for the analysis of biomarkers in the CSF (amyloid-β, tau); B) genetic analyses on peripheral blood: quantification of plasma progranulin and (according to the results) screening for mutations of the progranulin gene; apolipoprotein E genotyping.

Statistics. Cross-sectional analyses for inter-group comparisons (PPA groups, healthy controls) and longitudinal analyses for inter-group and intra-group comparisons (M0, M9, M18).

ELIGIBILITY:
Inclusion criteria A) Patients responding to current diagnostic criteria for Primary Progressive Aphasia

1. Language disorders without important impairments of other cognitive functions
2. Insidious onset and gradual progression

   * Diagnostic criteria for non fluent PPA
   * Non fluent language out-put
   * Phonemic paraphasias and/or agrammatism
   * Relative preservation of speech comprehension
   * Diagnostic criteria for fluent PPA
   * Fluent language out-put
   * Impairment of the access to word meanings leading to comprehension disorders and naming deficits
   * Associative agnosia and/or prosopagnosia may be present. This will allow for the inclusion of patients with multi-modal disorders of meaning (semantic dementia patients).
   * Diagnostic criteria for logopenic PPA
   * Speech out-put with frequent interruptions due to word finding deficits
   * Disorders of sentence comprehension and repetition due to impairment of working memory B) Patients at age of majority C) Patients having given informed and written consent

Exclusion criteria A) Cognitive criteria

* Aphasia severity rating scale of the BDAE < 3
* MMS < 20
* Severe disorders of executive functions, praxis or episodic memory B) MADRS ≥ 20 (major depression as defined by criteria of the DSM-IV-R) C) Patients whose mother tongue is not French D) Patients affected by of other neurological diseases than PPA or general diseases or physical problems that may impact on cognitive functioning E) Counter-indication for MRI or PET scanning (the lumbar puncture is optional / separated informed consent) F) MRI compatible with pathological processes other than PPA. A mild to moderate leucoaraiosis will not been considered as an exclusion criteria (only patients at stage > 2 will be excluded from the study) G) Non affiliation at the French healthcare system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2012-03; Primary Completion 2017-03 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Composite outcome mesure using multiple cognitive, imaging and biological parameters | D0
  Characterisation of the three PPA variants investigating 1) the cognitive features (psycholinguistic), 2) the anatomic/metabolic substrates (structural MRI, DTI-based tractography, functional connectivity fMRI-resting state, 18FDG-PET), and 3) the biologic aspects (CSF biomarkers [amyloid-β, tau], genetic screening for mutations in the progranulin gene, apolipoprotein E genotyping).
Composite outcome mesure using multiple cognitive, imaging and biological parameters | 9 months
  Characterisation of the three PPA variants investigating 1) the cognitive features (psycholinguistic), 2) the anatomic/metabolic substrates (structural MRI, DTI-based tractography, functional connectivity fMRI-resting state, 18FDG-PET), and 3) the biologic aspects (CSF biomarkers [amyloid-β, tau], genetic screening for mutations in the progranulin gene, apolipoprotein E genotyping).
Composite outcome mesure using multiple cognitive, imaging and biological parameters | 18 months
  Characterisation of the three PPA variants investigating 1) the cognitive features (psycholinguistic), 2) the anatomic/metabolic substrates (structural MRI, DTI-based tractography, functional connectivity fMRI-resting state, 18FDG-PET), and 3) the biologic aspects (CSF biomarkers [amyloid-β, tau], genetic screening for mutations in the progranulin gene, apolipoprotein E genotyping).

CONTACTS AND LOCATIONS:
Overall Officials: Marc Teichmann, MD, PhD, Principal Investigator — Assitance Publique-Hopitaux de Paris
Locations (1):
- Département de Neurologie - Centre des maladies neurologiques, cognitives et comportementales, France, France